CLINICAL TRIAL: NCT00969241
Title: The Effect of Periodontal Treatment on the Level of Free Radicals in the Saliva
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Dr. front the department of oral and maxillofacial surgery, the department of oral and maxillofacial surgery - poria madical center
Other Study IDs: 920090018-YR.ctil
Record Dates: First submitted 2009-08-30; First posted 2009-09-01 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2009-08

CONDITIONS: Periodontitis
Keywords: saliva; free-radicals; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will examine the relationship between free radicals in the saliva and periodontitis. 30 adults, 15 with periodontitis and 15 as a control group will give a sample of saliva before treatment and after treatment. The investigators will examine the free radicals in both groups.

DETAILED DESCRIPTION:
Periodontal disease is a chronic adult condition. Bacteria implicated in the etiology of this disease causes destruction of connective tissue and bone. As a result of stimulation by bacterial antigen PMN produces free radicals via respiratory burst as a part of host response to infection.

Free radicals can be defined as molecules or molecular fragments with an unpaired electron which imparts certain characteristics to the free radicals such as reactivity . Reactive free radicals are able to produce chemical modifications and to damage proteins, lipids, carbohydrates and nucleotides in the tissues.

ELIGIBILITY:
Inclusion Criteria:

* older than 18
* no medical problems

Exclusion Criteria:

* medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with periodontitis who visit the department and volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: eran front, Dr., Principal Investigator — department of oral and maxillofacial surgery
Locations (1):
- department of oral and maxillofacial surgery, Baruch Padeh Medical Center, Tieberia, Israel, Poria, Israel